CLINICAL TRIAL: NCT04075032
Title: Effect of a Pomegranate Extract on Metabolic and Inflammatory Markers, and the Gut Microbiota of Poly-medicated Metabolic Syndrome Patients
Brief Title: Pomegranate Consumption by Poly-medicated Metabolic Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital General Universitario Reina Sofía de Murcia (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AGL2015-64124-R(2)
Record Dates: First submitted 2019-08-22; First posted 2019-08-30 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; pomegranate; gut microbiota; polyphenol; polymedication; inflammation; obesity; diabetes; hypertension; hyperlipidemia; urolithins
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Obesity; Diabetes Mellitus; Hypertension; Hyperlipidemias | interventions — pomegranate fruit rind

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled and crossover trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pomegranate extract-1 (Experimental): Consumption of 2 daily capsules (900 mg pomegranate extract, PE) for 4 weeks
  Interventions: Dietary Supplement: Pomegranate extract
- Placebo-1 (Placebo Comparator): Consumption of 2 daily capsules (900 mg microcrystalline cellulose, PLA) for 4 weeks
  Interventions: Other: Placebo
- Placebo-2 (Placebo Comparator): Consumption of 2 daily capsules (900 mg microcrystalline cellulose, PLA) for 4 weeks. This arm is the previous PE-1 after crossover and one month of wash-out
  Interventions: Other: Placebo
- Pomegranate extract-2 (Experimental): Consumption of 2 daily capsules (900 mg pomegranate extract, PE) for 4 weeks. This arm is the previous PLA-1 after crossover and one month of wash-out.
  Interventions: Dietary Supplement: Pomegranate extract

INTERVENTIONS:
Dietary Supplement: Pomegranate extract — Pomegranate extract consumption (900 mg/day) for 4 weeks
  Arms: Pomegranate extract-1; Pomegranate extract-2
Other: Placebo — Placebo (microcrystalline cellulose) consumption (900 mg/day) for 4 weeks
  Arms: Placebo-1; Placebo-2

SUMMARY:
The objective is to evaluate whether the medication in polymedicated metabolic syndrome patients could determine the effects of a pomegranate extract on i) metabolic markers, ii) inflammatory markers, and iii) the modulation of the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >30 kg/m2 or waist circumference >94/80 cm (males/females) in European-Caucasians subjects, plus two of the following:
* Triglycerides >150 mg/dL or under treatment against hypertrigliceridemia.
* Fasting glucose ≥100 mg/dL
* Diagnosed type 2 diabetes mellitus
* HDL-cholesterol (mg/dl) <40/50 (males/females) or under treatment against low HDLc values.
* Systolic blood pressure >130 mmHg o diastolic blood pressure >85 mmHg, or under anti-hypertensive drug treatment.

Exclusion Criteria:

* Age under 18 years
* Pregnancy or breastfeeding
* Antibiotic treatment within one month before inclusion in the trial
* Pomegranate allergy or intolerance (known or suspected)
* Chronic intestinal inflammatory diseases (ulcerative colitis, Crohn's disease, etc.)
* Malignancies
* Consumption of botanicals or dietary supplements within one month before the inclusion and during the trial.
* Consumption of ellagitannin-rich sources within one week before the inclusion and during the trial (pomegranate, walnuts, strawberries, raspberries, tea, blackberries and oak-aged wine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change (1 log units) of Bacteroidetes per gram of feces | Change from baseline at 30 days vs placebo
  Modulation of gut microbiota (decrease Firmicutes to Bacteroidetes ratio)

SECONDARY OUTCOMES:
Change (10%) of circulating levels of lipopolysaccharide binding protein (LBP) | Changes from baseline at 30 days vs placebo
  Evaluation of metabolic endotoxemia
Change (10%) of ghrelin, TNF-α, GLP-1, IL-6, PYY, resistin, HGF, MCP-1, C-Peptide, and BDNF (pg/mL). | Changes from baseline at 30 days vs placebo
  Determination of metabolic and inflammatory markers in serum samples.
Change (10%) of PAI-1, adiponectin, RBP4, and leptin (ug/mL). | Changes from baseline at 30 days vs placebo
  Determination of fibrinolytic, inflammatory and metabolic markers in serum samples
Change (10%) of ICAM-1, VCAM-1, and P-selectin (ng/mL) | Changes from baseline at 30 days vs placebo
  Measurement of cell adhesion molecules in serum samples
Change (10%) of blood glucose, total cholesterol, LDLc and HDLc concentrations (mg/dL) | Changes from baseline at 30 days vs placebo
  Measurement of serobiochemical variables (blood glucose and lipids levels) in serum samples
Evaluation of genotype frequencies for 60 single nucleotide polymorphisms (SNPs) related to the incidence of obesity, metabolism, diabetes and cardiovascular diseases | Baseline values at inclusion
  SNP genotyping of patients (DNA extracted from whole blood)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Espín, PhD, Principal Investigator — Spanish National Research Council (CSIC)
Locations (1):
- Spanish National Research Council (CSIC), Murcia, Spain